CLINICAL TRIAL: NCT01097798
Title: Multicenter, Randomized, Double-blind Trial to Evaluate the Efficacy and Safety Aliviador Compared to Gelol in the Relief in Patients With Contusons, Sprains,Trauma and Muscle Injury.
Brief Title: To Evaluate the Efficacy and Safety Aliviador Compared to Gelol in Patients With Contusions, Sprains, Trauma and Muscle Injury.
Acronym: LBB-ALI-01/09
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratorio Brasileiro de Biologia (Other)
Responsible Party: Maria Lygia Bezerra, Laboratório Brasileiro de Biologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBB-ALI-01/09
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-02

CONDITIONS: Contusions; Sprains; Trauma; Muscle Injury; Myalgia; Myofascial Pain; Tendinitis
Keywords: muscle injury
MeSH Terms: conditions — Contusions; Sprains and Strains; Wounds and Injuries; Myalgia; Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliviador (Experimental)
  Interventions: Drug: Aliviador
- Gelol (Active Comparator)
  Interventions: Drug: Gelol

INTERVENTIONS:
Drug: Aliviador — The study medication should be applied regimen of 8/8 hours over 2 days.
  Arms: Aliviador
Drug: Gelol — The study medication should be applied regimen of 8/8 hours over 2 days.
  Arms: Gelol

SUMMARY:
Multicenter, randomized, double-blind trial, to evaluate the efficacy and safety Aliviador compared to Gelol in the relief of signs and symptoms in patients with contusions, sprains, trauma and muscle injury start with less than 24 hours or patients of myalgia, myofascial pain and tendinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, of any race, aged over 12 years.
* Ability to read, understand and sign the IC, in the case of minors consent of responsible;
* Clinical diagnosis of bruises, sprains, trauma, muscle damage occurred in less than 24 hours or muscle pain, myofascial pain or tendinitis.
* Patients able to understand and maintain the clinical protocol.

Exclusion Criteria:

* Known hypersensitivity to components of the formulas of both the drug test as the comparator.
* Known hypersensitivity to paracetamol.
* Location of the lesion with skin wound or irritated.
* Liver or kidney disease known.
* Pregnant or lactating women.
* Patients who require surgery or immobilization.
* Patients with fractures or rupture of the ligaments.
* Patients using anticoagulants.
* Patients with severe concomitant systemic diseases, such as cancer, diabetes, or acquired heart disease, hematological diseases, seizure disorders, autoimmune diseases, renal failure, severe infections, hormonal disorders and pulmonary disorders.
* History of alcoholism or illicit drug use;
* Use of NSAIDs, corticosteroids or venoterápicos, topics or any other form of administration.
* Conditions in the opinion of the researcher make the patient unsuitable to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy in reducing signs and symptoms Aliviador compared to Gelol. | two days
  To evaluate the efficacy in reducing signs and symptoms Aliviador compared to Gelol in patients with contusions, sprains, muscle injury and trauma, starting less than 24 hours or patients with muscle pain, myofascial pain and tendinitis.

SECONDARY OUTCOMES:
To evaluate the tolerability use Aliviador compared to Gelol. | two days
  To evaluete the tolerability use Aliviador compared to Gelol in patients with contusions, sprains, muscle injury and traumas starting less than 24 hours or patients with myalgia, myofascial pain and tendinitis.

CONTACTS AND LOCATIONS:
Overall Officials: Abel Pereira Junior, investigator, Principal Investigator — Faculdade de Medicina do ABC; Gilberto de Castro Brandão, investigator, Principal Investigator — Clínica Perdizes; Paulo Faria, investigator, Principal Investigator — S.C. Corinthians Paulista
Locations (3):
- Brazil (3):
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Clínica Perdizes, São Paulo, São Paulo
  - S.C. Corinthians Paulista, São Paulo, São Paulo